CLINICAL TRIAL: NCT04793659
Title: A Phase 2a Combined Open-Label and Double-Blind, Placebo-Controlled Crossover Study Assessing the Effectiveness, Safety, and Tolerability of Oral Fasudil in Subjects With Dementia and Wandering Behaviors of Elopement and/or Getting Lost
Brief Title: Fasudil fOr redUcing elopemeNt and Spatial Disorientation
Acronym: FOUND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Woolsey Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WP-0512-001
Record Dates: First submitted 2021-02-11; First posted 2021-03-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Dementia
Keywords: Wandering Behavior; Dementia; Fasudil
MeSH Terms: conditions — Dementia; Wandering Behavior | interventions — fasudil

STUDY DESIGN:
Intervention Model Description: Combined Open-Label and Double-Blind, Placebo-Controlled Crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Periods 1 and 2 of the open-label phase will be unblinded.
  Periods 3 and 4 are double-blind crossover phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Fasudil 90 mg/day (Experimental): Subjects will receive a daily dose of 90 mg Fasudil for 42 days (open-label period 1). After Period 1 is complete, if the subject is a responder to Fasudil 90 mg/day, they will be randomized to either Fasudil 90 mg/day or a placebo for 6 weeks (double-blind period 1), then crossover to the other arm for 6 weeks (double-blind period 2).
  Interventions: Drug: Oral Fasudil 90 mg/day; Drug: Oral Placebo
- Oral Fasudil 180 mg/day (Experimental): If the subject is a not a responder in the open-label period 1 but tolerated Fasudil 90 mg/day, they will be escalated to Fasudil 180 mg/day (open-label period 2) for 42 days. If the subject is a responder to Fasudil 180 mg/day, they are randomized to either Fasudil 180 mg/day for 42 days or a placebo (double-blind period 1), then crossover to the other arm for 6 weeks (double-blind period 2).
  Interventions: Drug: Oral Fasudil 180 mg/day; Drug: Oral Placebo
- Oral Placebo (Placebo Comparator): Placebo comparator arm to investigational drug (Fasudil 90 mg/day or 180 mg/day).
  Interventions: Drug: Oral Fasudil 90 mg/day; Drug: Oral Fasudil 180 mg/day; Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Fasudil 90 mg/day — Oral tablet
  Arms: Oral Fasudil 90 mg/day; Oral Placebo
Drug: Oral Fasudil 180 mg/day — Oral tablet
  Arms: Oral Fasudil 180 mg/day; Oral Placebo
Drug: Oral Placebo — Oral tablet

SUMMARY:
Fasudil, a Rho kinase inhibitor, is believed to reduce wandering behaviors of elopement and getting lost by improving spatial memory and navigation through improvements in hippocampal blood flow. Fasudil is non-sedating.

The aim of the study is to assess the effectiveness of oral fasudil in reducing wandering behaviors of elopement and/or getting lost in subjects with dementia. In addition, effects on wandering behaviors of excess movement and pacing, cognition, memory, neuropsychiatric symptomatology, caregiver/nursing staff burden, and the safety and tolerability of fasudil treatment will be assessed.

DETAILED DESCRIPTION:
The study population will consist of subjects with dementia and wandering behaviors of elopement and/or getting lost. While it is anticipated that most participants will be residing at home (with caregiver support), subjects may live in another setting such as a group home, an assisted living unit, or in a long-term care facility, provided that a caregiver, formal or informal, has sufficient contact with the subject to permit accurate completion of the necessary assessments.

Enrolled subjects will enter the Open-Label Phase and receive treatment with fasudil 90 mg/day (30 mg three times daily [tid]) for 6 weeks in Open-Label Period 1. Responders (i.e., subjects who improve 2 points or more on the GIW) will proceed to the Double-Blind Phase. Subjects in whom fasudil is well-tolerated (i.e. subjects with ≤ 2 drug-related AEs of mild intensity, no drug-related AEs of greater than mild intensity, and creatinine level of < 1.5 mg/dL at all times during the period) and who do not respond will enter Open-Label Period 2, and be dosed with fasudil 180 mg/day (60 mg tid) for 6 weeks. Responders will proceed to the Double-Blind Phase and non-responders will move to the final post-treatment visit. In the Double-Blind Phase, subjects will receive treatment with either placebo or the dose they responded to in the Open-Label Phase (90 mg/day or 180 mg/day) for 6 weeks (Double-Blind Period 1), following which treatment assignment will be crossed over for 6 weeks (Double-Blind Period 2). A final post-treatment visit will occur 14 days after the last dose of study drug. Visits may be performed by qualified healthcare professionals at home or other care setting, or at a doctor's office/clinic. Interviews may be performed by telephone and/or telemedicine as appropriate.

Study Endpoints:

Primary:

• The Global Impression of Wandering (GIW)

Secondary:

* Weekly Wandering Report - Community Version (WWR-C)
* The Revised Algase Wandering Scale - Community Version (RAWS-CV)
* The Mini Mental State Examination (MMSE)
* The Neuropsychiatric Inventory-Questionnaire (NPI-Q)
* The Cohen-Mansfield Agitation Inventory - Community Version (CMAI-C)
* The Center for Neurological Study-Lability Scale (CNS-LS)
* The Zarit Burden Interview (ZBI)
* Safety
* Tolerability

ELIGIBILITY:
Inclusion Criteria:

1. 50 to 90 years of age (inclusive).
2. Diagnosis of dementia of any etiology.
3. MMSE 9-24 (inclusive).
4. Presence of one or both of the following wandering behaviors that in the opinion of the investigator, in consultation with caregiver, is at least of moderate severity (defined as clearly a wanderer, and this causes some distress or difficulty for both the subject and caregiver):

   1. Elopes or attempts to elope AND/OR
   2. Gets lost or is unable to locate a specific place.
5. Independently ambulatory with or without assistive devices (such as canes or walkers). Subjects must not require assistance to transfer out of bed or a chair.
6. Subject has a caregiver who has more than 10 hours/week of contact with the subject, is fluent and literate in English and is willing to accept responsibility for supervising the treatment (e.g., administering study drug) and assessing the condition of the subject throughout the study in accordance with all protocol requirements.
7. Consent obtained from the participant/legally authorized representative (LAR) in accordance with local regulations.

Exclusion Criteria:

1. Expected change in medication that could interfere with the study or free movement of the subject.
2. Serum creatinine ≥ 1.5 mg/dL.
3. ALT and/or alkaline aminotransferase (AST) ≥ 2 X and/or alkaline phosphatase (ALP) ≥ 1.5 upper limit of normal.
4. Blood pressure < 90/60.
5. On more than one of the following drug classes: long-acting nitrates, beta-blockers, or calcium channel blockers.
6. Any severe comorbidity that in the opinion of the Investigator would disallow safe participation in the trial.
7. Women of child-bearing potential; females must be postmenopausal or surgically sterilized.
8. Suicidal ideation per the Columbia-Suicide Severity Rating Scale (C-SSRS) that in the opinion of the PI would pose a safety risk or interfere with the appropriate interpretation of study data.
9. Planned change in the current living setting during the study.
10. History within the last year of either two or more falls leading to clinically significant injuries or one or more fall leading to hospitalization, and/or evidence of orthostatic hypotension.
11. Participation in another investigational drug study within 30 days before start of Open-Label period.
12. Subjects who, in the opinion of the investigator, are not suitable for the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Global Impression of Wandering (GIW) after oral Fasudil vs placebo in the Double-Blind Phase | Week 6 and Week 12 of the Double-Blind period
  The GIW is a variant of the 7-point Clinical Global Impression-Severity (CGI-S) scale and is used in FOUND specifically to obtain the investigator's overall assessment of severity of the subject's wandering behavior.

SECONDARY OUTCOMES:
Change in Weekly Wandering Report - Community Version (WWR-C) | Weekly during the 12 weeks of the Double-Blind period
  The WWR-C is composed of targeted questions related to excess walking, spontaneous pacing, elopement, and wayfinding; it is designed to be assessed on a weekly basis by caregivers about subjects for whom they care. The WWR-C asks the caregiver to rate the subject's behavior for the previous week.
Change in the Revised Algase Wandering Scale - Community Version (RAWS-CV) | Week 6 and Week 12 of the Double-Blind period
  The RAWS-CV is a 40-item tool with 6 subscales to assess wandering behaviors (eloping behaviors, negative outcomes, mealtime impulsivity, persistent walking, repetitive walking, and spatial disorientation), and a total score scale.
Change in Mini Mental State Examination (MMSE) | Week 6 and Week 12 of the Double-Blind period
  The MMSE is a 30-point questionnaire that is used to measure cognitive impairment.
Change in Neuropsychiatric Inventory-Questionnaire (NPI-Q) | Week 6 and Week 12 of the Double-Blind period
  The NPI-Q provides an assessment of dementia-related emotional behavioral symptomatology in routine clinical practice settings. Caregiver distress is also assessed.
  The NPI-Q asks the assessor to rate the previous 30 days. At the Final Visit, the assessor will rate the NPI-Q for the 2-week period following the final dose. The scale is completed by the caregiver without input from the subject. All reasonable efforts should be made to ensure each NPI-Q for an individual subject is completed by the same caregiver to minimize inter-rater variability.
Cohen-Mansfield Agitation Inventory - Community Version (CMAI-C) | Week 6 and Week 12 of the Double-Blind period
  The CMAI-C is a 37-item scale to systematically assess agitation.
Center for Neurological Study-Lability Scale (CNS-LS) | Week 6 and Week 12 of the Double-Blind period
  The CNS-LS is a 7-item questionnaire to assess perceived frequency of pseudobulbar affect episodes.
Zarit Burden Interview (ZBI) | Week 6 and Week 12 of the Double-Blind period
  The ZBI is a 22-item scale to assess caregiver burden.
Adverse Events (AEs) | Through study completion, up to 26 weeks
Serious Adverse Events (SAEs) | Through study completion, up to 26 weeks
Change in blood pressure | Through study completion, up to 26 weeks
Change in blood parameters | Through study completion, up to 26 weeks
  Hematology: white blood cell count, hemoglobin, hematocrit, platelet count
Change in blood chemistry | Through study completion, up to 26 weeks
  Blood chemistry: glucose, sodium, potassium, bicarbonate, blood urea nitrogen, creatinine, cystatin c
Change in liver function | Through study completion, up to 26 weeks
  Liver function tests: albumin, total bilirubin, direct bilirubin, ALP, AST, ALT, gamma glutamyl transferase, lactate dehydrogenase
Change in urine contents | Through study completion, up to 26 weeks
  Urinalysis (occult blood, protein)
Change in heart rhythm | Through study completion, up to 26 weeks
  12-lead Electrocardiogram (ECG) will be used to obtain a record of cardiac activity
Change in body weight | Through study completion, up to 26 weeks
Change in body temperature | Through study completion, up to 26 weeks
Change in respiratory rate | Through study completion, up to 26 weeks
Columbia Suicide Severity Rating Scale (C-SSRS) | Through study completion, up to 26 weeks
  The C-SSRS is an assessment used to identify immediate risk of suicide, and is completed following the patient interview, review of medical record(s) and/or consultation with family members and/or other professionals. While the C-SSRS is a detailed interview, the full interview is needed only if the initial screening questions about suicidal ideation and behavior are positive.
  In subjects with severe cognitive impairment, i.e., so substantial as to interfere with an understanding of the concept of suicide, the C-SSRS may be omitted.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Accel Research Sites, Lakeland, Florida
  - Lakes Research, LLC., Miami Lakes, Florida
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Re:Cognition Health, Fairfax, Virginia
- Australia (5):
  - Modbury Hospital, Modbury, South Australia
  - Barwon Geriatrics, Geelong, Victoria
  - GV Health, Shepparton, Victoria
  - Northeast Health Wangaratta, Wangaratta, Victoria
  - Neurodegenerative Disorders Research, West Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No